CLINICAL TRIAL: NCT01017640
Title: ABT-888 as Monotherapy and in Combination With Mitomycin C in Patients With Solid Tumors With Deficiency in Homologous Recombination Repair
Brief Title: Veliparib With or Without Mitomycin C in Treating Patients With Metastatic, Unresectable, or Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01473; NCI-2012-01473 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU-09100; OSU# 09100; 2009C0069; 09100; NCI 8472; CDR0000656393; OSU 09100 (Other: Ohio State University Comprehensive Cancer Center); 8472 (Other: CTEP); N01CM00070 (NIH); N01CM62207 (NIH); P30CA016058 (NIH)
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Solid Neoplasm
MeSH Terms: interventions — Mitomycin; Mitozytrex; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (veliparib) (Experimental): Patients receive veliparib PO BID in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Veliparib
- Arm II (veliparib and mitomycin C) (Experimental): Patients receive veliparib PO BID on days 1-7, 1-14, or 1-21. Patients also receive mitomycin C IV over 10-20 minutes on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Mitomycin; Drug: Veliparib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mitomycin — Given IV
  Other Names: Ametycine; MITO; MITO-C; Mito-Medac; Mitocin; Mitocin-C; Mitolem; MITOMYCIN C; Mitomycin-C; Mitomycin-X; Mitomycine C; Mitosol; Mitozytrex; Mutamycin; Mutamycine; NCI-C04706
  Arms: Arm II (veliparib and mitomycin C)
Drug: Veliparib — Given PO
  Other Names: ABT-888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I trial studies the side effects and best dose of veliparib when given with or without mitomycin C in treating patients with solid tumors that have spread to other places in the body, cannot be removed by surgery or have come back. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as mitomycin C, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving veliparib together with mitomycin C may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To screen cancer patients across different histological sites to identify those with functional defects in the Fanconi anemia (FA) pathway in their tumors.

II. To establish the safety and practicality of treating patients with FA deficient tumors with the poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitor ABT-888 (veliparib) as protracted monotherapy.

III. To establish the safety and practicality of treating patients with FA deficient tumors with the combination of mitomycin C (MMC) and ABT-888.

IV. To select a dose of ABT-888 protracted monotherapy and a dose-schedule of the combination of mitomycin C and ABT-888 in patients with FA deficient tumors for phase 2 trials.

SECONDARY OBJECTIVES:

I. To evaluate for germ-line FA repair deficiency and BRCA mutations in peripheral blood mononuclear (PBMC) in patients receiving ABT-888 treatment.

II. To evaluate in PBMC samples for foci produced by the histone variant gamma-H2A histone family, member X (H2AX) in patients receiving mitomycin C with or without ABT-888 in order to assess any possible effect of ABT-888 in the cellular sensing and processing of mitomycin C-induced deoxyribonucleic acid (DNA) double strand breaks.

III. Quantify the number of patients with antitumor responses.

OUTLINE: This is a dose-escalation study of veliparib. Patients are assigned to 1 of 2 treatment arms.

ARM I: Patients receive veliparib orally (PO) twice daily (BID) in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive veliparib PO BID on days 1-7, 1-14, or 1-21. Patients also receive mitomycin C intravenously (IV) over 10-20 minutes on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed solid malignancy that is metastatic, or unresectable, or recurrent, for which no curative or standard of care exist, or this standard of care is no longer effective
* Tumors have been shown to be deficient for the FA pathway, based on Fanconi anemia triple stain immunofluorescence (FATSI) screening
* Patients will be consented to have their existing, or about to be obtained, paraffin embedded tumor tissue screened for FA deficiency; screening will be performed on an ongoing basis on the breast, thoracic, gastrointestinal (GI), Georgetown University (GU), and gynecologic (GYN) Ohio State University (OSU) clinics, anteceding and concurrently with the clinical trial; it will continue until the numbers of patients required for the clinical trial are identified and enrolled; based on the estimation from our preliminary data of 15 to 30% of patients, depending on the primary organ site, having tumors deficient for the FA pathway we will need to screen around 300 patients' samples to identify 40-50 patients; none of the eligibility criteria defined above or below will need to be met for the screening portion, since FA deficient patients identified by screening may meet eligibility criteria for the clinical trial at a later time; (e.g., patient is undergoing standard of care treatment at the time of the screening); separate written consents for screening and for the clinical trial will be obtained from patients
* Up to two chemotherapy regimens for metastatic disease are allowed; in addition, prior adjuvant/neo-adjuvant chemotherapy, hormonal therapy, molecular targeted therapy or estrogen receptor B (Erb) inhibitor treatments (e.g., erlotinib, Herceptin, sorafenib, sunitinib) will be allowed and will not count towards eligibility; at least 4 weeks must elapse since prior chemotherapy or radiation therapy (two weeks for erlotinib, hormonal therapy, or limited field palliative radiation to bone, brain, or radiosurgery), 6 weeks if the last regimen included nitrosoureas or mitomycin C; previous use of mitomycin C would be restricted to topical applications (bladder cancer) or chemoembolization (e.g., liver tumors)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Hemoglobin >= 9 g/dL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limit
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Patients should be able to swallow capsules
* EXPANSION COHORT:

  * Diagnosis of colorectal malignancy
  * Absence of Fanconi anemia, complementation group D2 (FANCD2) foci by FATSI screening
  * Presence of biopsiable lesion by imaging
  * Consent to a baseline (prior to treatment) tumor biopsy and for a repeat biopsy at the time of progression on the event that an antitumor response is demonstrated on the MMC-ABT-888 regimen
  * Same eligibility as above, except that they will have no limitations related prior number of chemotherapy regimens given; patients could have received prior treatment with PARP inhibitors if used as single agent

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Patients with known central nervous system (CNS) metastases (unless previously resected or irradiated and not clinically active); patients with CNS metastases must be stable after therapy for > 3 months and off steroid treatment prior to study enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition as ABT-888 or Mitomycin C
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patients with active seizure or a history of seizures
* Patients previously treated with PARP inhibitors; with the exception of patients enrolled on Arm 2 who may have had prior treatment with PARP inhibitors as monotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Ability to safely deliver the combination of mitomycin C and veliparib | Up to 12 weeks post-treatment
Ability to safely deliver veliparib in a continuous dose as monotherapy | Up to 12 weeks post-treatment
Feasibility of screening for FA deficiency across different tumor types, defined as adequate number of patients deficient on this pathway | Up to 12 weeks post-treatment
Selection of a dose schedule of the combination of mitomycin C and veliparib for phase II trials | Up to 12 weeks post-treatment
Selection of a dose schedule of veliparib monotherapy for phase II trials | Up to 12 weeks post-treatment

SECONDARY OUTCOMES:
BRCA mutations | Baseline
  Descriptive statistics will be provided: proportions for categorical variables; mean and standard deviation for the continuous variables.
FancD2 foci formation in peripheral blood mononuclear cells | Up to week 5
  Descriptive statistics will be provided: proportions for categorical variables; mean and standard deviation for the continuous variables.
Foci produced by the histone variant gamma-H2AX | Up to week 5
  Descriptive statistics will be provided: proportions for categorical variables; mean and standard deviation for the continuous variables.
Tumor shrinkage as assessed by radiological means | Up to 12 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Mikhail, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Georgetown Cancer Treatment Center, Georgetown, Kentucky
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio